CLINICAL TRIAL: NCT03532945
Title: A Long-term Follow-up Study to Evaluate the Efficacy and Safety for the Patients With Bioactive Glass-ceramic Intervertebral Spacer (Novomax) in Posterior Lumbar Interbody Fusion: Comparison With a Titanium Cage
Brief Title: A Follow-up Study to Evaluate the Efficacy and Safety of Novomax in Posterior Lumbar Interbody Fusion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BioAlpha Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B1504
Record Dates: First submitted 2018-05-02; First posted 2018-05-22 (Actual); Last update posted 2018-05-22 (Actual); Status verified 2018-05

CONDITIONS: Degenerative Lumbar Spinal Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bioactive Glass-Ceramic Spacer (Experimental): The one-level Posterior Lumbar Interbody Fusion(PLIF) surgery will be carried out with Novomax, which is the bioactive glass ceramic intervertebral spacer.
  Interventions: Device: Bioactive Glass-Ceramic Spacer
- Titanium cage (Active Comparator): The one-level Posterior Lumbar Interbody Fusion(PLIF) surgery will be carried out with titanium cage.
  Interventions: Device: Titanium cage

INTERVENTIONS:
Device: Bioactive Glass-Ceramic Spacer
  Other Names: Novomax
  Arms: Bioactive Glass-Ceramic Spacer
Device: Titanium cage
  Arms: Titanium cage

SUMMARY:
This is a long-term follow-up study for more than 3 years to evaluate the efficacy and safety of bioactive glass-ceramic intervertebral spacer (Novomax) in posterior lumbar interbody fusion.

DETAILED DESCRIPTION:
During one-level PLIF, bioactive glass-ceramic intervertebral spacer (Novomax) and titanium cage were inserted in the experimental group and control group, respectively. Bone fusion by simple radiography had angular deformity of less than 3 degrees and a potential of less than 3 mm in flexion extension radiographs, and thin-section CT (<2 mm) was used to determine the combination between the vertebral endplate and the autogenous bone or bioactive glass-ceramic intervertebral spacer (Novomax) in the cage without any gaps or the part connected to bony trabecula as fusion, and both groups will be compared.

ELIGIBILITY:
Inclusion Criteria:

[In Interventional Study]

* Subjects who required between L1 and S1 among those who required an extensive laminectomy or facetectomy to correct severe disc extrusion or severe spinal stenosis or those who required PLIF due to grade I or II spondylolisthesis

[In Long-term Follow-up Study]

* Subjects who are treated with bioactive glass ceramic intervertebral spacer or titanium cage in one-level PLIF surgery

Exclusion Criteria:

[In Interventional Study]

* Subjects with average T-scores of L1-L4 at <-3.0 in DEXA bone density tests
* Subjects who are pregnant or breast-feeding
* Subjects with a history of malignant tumor or malignant diseases (but the cases of cured disease with no relapse for the past 5 years were included in the present study)
* Subjects with abnormal blood potassium and phosphorus levels
* Subjects who are considered not suitable for the study by significant disease(liver disease, kidney disease, respiratory disease, metabolic disease, or psychological disease)
* Subjects who are not able to comply with the study requirements
* Subjects who are considered not suitable for the study by the investigator

[In Long-term Follow-up Study]

* Subjects who are not able to comply with the study requirements
* Subjects who are considered not suitable for the study by the investigator

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2010-10-28 (Actual); Primary Completion 2013-09-13 (Actual); Study Completion 2016-04-07 (Actual)

PRIMARY OUTCOMES:
Bone fusion with radiographs (X-ray) | for 36 months after surgery
  Evaluation of bone fusion between bone substitutes and vertebral endplates with X-ray for 36 months(or more than 36 months) after PLIF surgery.

SECONDARY OUTCOMES:
Bone fusion with 3-dimensional computed tomography(CT) | for 36 months after surgery
  Evaluation of bone fusion between bone substitutes and vertebral endplates with 3-dimensional CT for 36 months(or more than 36 months) after PLIF surgery.
The Oswestry Disability Index(ODI) assessment | for 36 months after surgery
  Evaluation of the Oswestry disability index questionnaire survey for 36 months(or more than 36 months) after PLIF surgery.
The SF(Short Form)-36 questionnaire assessment | for 36 months after surgery
  Evaluation of the SF(Short Form)-36 questionnaire survey for 36 months(or more than 36 months) after PLIF surgery.
VAS for target site | for 36 months after surgery
  Evaluation of target site pain using the visual analogue scale (VAS) for 36 months(or more than 36 months) after PLIF surgery.
1.Number of Participants with Adverse Events as a Measure of Safety and Tolerability | for 36 months after surgery
  Evaluation of AE

CONTACTS AND LOCATIONS:
Overall Officials: Bong-Soon Chang, MD. PhD., Principal Investigator — Seoul National University Hospital; Ki Hyoung Koo, MD. PhD., Principal Investigator — DongGuk University; Ho-Joong Kim, MD. PhD., Principal Investigator — Seoul National University Bundang Hospital; Jae Hyup Lee, MD. PhD., Principal Investigator — SMG-SNU Boramae Medical Center

IPD SHARING:
Plan to Share IPD: Undecided